CLINICAL TRIAL: NCT02931747
Title: Effect of Bacopa Monnieri on Working Memory and Cognitive Processing in Student
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Khon Kaen University (Other)
Collaborators: Government Pharmaceutical Organization (Unknown)
Responsible Party: Principal Investigator, Jintanaporn Wattanathorn, Associated Professor Doctor, Khon Kaen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HE581418
Record Dates: First submitted 2016-10-08; First posted 2016-10-13 (Estimated); Last update posted 2017-08-18 (Actual); Status verified 2017-08

CONDITIONS: Healthy
Keywords: Bacopa Monnieri; Working memory; Cognitive processing; Student

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Subjects are received the pill of placebo which has same color, shape and smell like the Bacopa Monnieri once daily for 16 weeks.
  Interventions: Dietary Supplement: Placebo
- Bacopa Monnieri 300 mg/day (Active Comparator): Subjects are received the pill of Bacopa Monnieri at the dose of 300 mg/day once daily for 16 weeks
  Interventions: Dietary Supplement: Bacopa Monnieri 300 mg/day
- Bacopa Monnieri 600 mg/day (Active Comparator): Subjects are received the pill of Bacopa Monnieri at the dose of 600 mg/day once daily for 16 weeks
  Interventions: Dietary Supplement: Bacopa Monnieri 600 mg/day

INTERVENTIONS:
Dietary Supplement: Placebo — Subjects are received Placebo once daily for 16 weeks.
  Arms: Placebo
Dietary Supplement: Bacopa Monnieri 300 mg/day — Subjects are received Bacopa Monnieri at the dose of 300 mg/day once daily for 16 weeks.
  Arms: Bacopa Monnieri 300 mg/day
Dietary Supplement: Bacopa Monnieri 600 mg/day — Subjects are received Bacopa Monnieri at the dose of 600 mg/day once daily for 16 weeks.
  Arms: Bacopa Monnieri 600 mg/day

SUMMARY:
The purpose of this study is to determine the effect of Bacopa Monnieri on working memory and cognitive processing in student.

DETAILED DESCRIPTION:
Learning and working memory are two of the key role for studying and work successful for student particular the high school student who study hard and preparing themselves for the graduate study. The consumption of brain booster product or functional food for improving memory has gained much attention. It has been reported that Bacopa Monnieri could improve learning and working memory in elderly subject by improving the N100 and P300 event related potential. Therefore, Bacopa Monnieri might be the potential product for improving the learning and working memory in student particular high school student.

ELIGIBILITY:
Inclusion Criteria:

* Healthy student subject aged between 15-18 years old who studying in the school within Khon Kaen province.
* Body mass index is between 18.5-24.9

Exclusion Criteria:

* Subjects who are diagnosed with one of the following: cardiovascular diseases, respiratory disease, neuropsychological diseases, head injury, diabetes mellitus, liver disease, cancer, autoimmune disease and hematological disorder are excluded.
* Subjects who take any medicine or nutraceuticals or hormone that effect on central nervous system are excluded.
* Alcohol addict or smoking addiction (more than 10 pieces/day)
* Athlete or subjects who have a regular exercise more than 3 times/week
* Subjects who don't follow the instruction during the trial
* Subjects who are participating the other project.

Ages: 15 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 75 (Actual)
Dates: Start 2016-07; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Cognitive processing using the latency of P300 wave | 4 months
  The latency of P300 wave was measured and expressed as millisecond.
Cognitive processing using the amplitude of P300 wave | 4 months
  The amplitude of P300 wave was measured and expressed as micro-volt.
Attention using the latency of N100 wave | 4 months
  The latency of N100 wave was measured and expressed as millisecond.
Attention using the amplitude of N100 wave | 4 months
  The amplitude of N100 wave was measured and expressed as micro-volt.

SECONDARY OUTCOMES:
Accuracy of working memory using computerized battery test | 4 months
  The accuracy of working memory was determined and expressed as percentage.
Speed of working memory using computerized battery test | 4 months
  The speed of working memory was determined and expressed as millisecond.
Assessment of psychiatric symptoms using the symptom check list 90 (SCL-90) | 4 months
Assessment of mood scale using Bond-Lader visual analogue scales | 4 months
Acetylcholinesterase activity in serum | 4 months
Monoamine oxidase activity in serum | 4 months
Glutamic acid decarboxylase (GAD) activity in serum | 4 months
Gamma-aminobutyric acid (GABA)-transaminase in serum | 4 months
Malondialdehyde level in serum | 4 months
Activity of superoxide dismutase in serum | 4 month
Activity of catalase in serum | 4 month
Activity of glutathione peroxidase in serum | 4 month
Consumption safety of Bacopa Monnieri using electrocardiogram (EKG) | 4 month
Consumption safety of Bacopa Monnieri using hematological values . | 4 month
  The hematological values including red blood cell, white blood cell, hematocrit and platelet were determined and the data was expressed as number of subject presented with abnormal hematological value.
Consumption safety of Bacopa Monnieri using blood chemistry | 4 month
  The blood chemistry values including renal function test, liver function test, lipid profile, electrolytes and glucose were determined and the data was expressed as number of subject presented with abnormal blood chemistry value.
Consumption safety of Bacopa Monnieri using blood pressure measurement | 4 month

CONTACTS AND LOCATIONS:
Locations (1):
- Jitanaporn Wattanathorn, Khon Kaen, Thailand

IPD SHARING:
Plan to Share IPD: No